CLINICAL TRIAL: NCT01387854
Title: A Re-Survey Study of Patients With MPS VI (Maroteaux-Lamy Syndrome) Who Previously Participated in ASB-00-02
Brief Title: Observational Study of Patients With Mucopolysaccharidosis (MPS) VI Who Previously Participated in ASB-00-02
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: ASB-00-03
Record Dates: First submitted 2011-06-29; First posted 2011-07-06 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: MPS VI
MeSH Terms: conditions — Mucopolysaccharidosis VI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
There is limited information on the long-term effects of treating patients with MPS VI with Naglazyme® and limited data on the natural history of treated and untreated MPS VI patients. The Re-survey Study ASB-00-03 will assist in understanding the effects of long-term Naglazyme treatment and the natural history of the MPS VI patient population.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent, or in the case of patients under the age of 16 years, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Previously participated in Survey Study ASB-00-02, and met the criteria of a MPS VI diagnosis.
* Willing to perform all study assessments and procedures as physically possible.

Exclusion Criteria:

* Concurrent disease or condition that would interfere with study participation or safety.
* Any condition that, in the view of the Investigator would place the patient at high risk of not completing the study.
* Concurrent enrollment and randomization into a clinical study of MPS VI treatment. Patients enrolled in the BioMarin MPS VI Clinical Surveillance Program may be enrolled in the Re-survey Study ASB-00-03.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with MPS VI who previously participated in ASB-00-02
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-06; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Linear Comparison of assessments completed for Survey Study ASB-00-02 and and Re-Survey StudyASB-00-03 | Variable dependent on date of assessment performed fo rthe Survey STudy ASB-00-02
  This study is designed to be performed in a similar manner to the Survey Study ASB-00-02. Similar assessments will be performed in order to make linear comparisons in outcomes over a long-term period.

CONTACTS AND LOCATIONS:
Locations (7):
- Children's Hospital and Research Center, Oakland, California, United States
- Women's and Children's hospital, North Adelaide, Australia
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil
- Hôpital Femme Mère Enfant, Lyon, Lyon, France
- Prof Michael Beck, Mainz, Mainz, Germany
- Al. Prof Hernani Monteiro, Porto, Porto District, Portugal
- Manchester Academic Health Sciences Centre, Manchester, Manchester, United Kingdom

REFERENCES:
- [Derived] Giugliani R, Lampe C, Guffon N, Ketteridge D, Leao-Teles E, Wraith JE, Jones SA, Piscia-Nichols C, Lin P, Quartel A, Harmatz P. Natural history and galsulfase treatment in mucopolysaccharidosis VI (MPS VI, Maroteaux-Lamy syndrome)--10-year follow-up of patients who previously participated in an MPS VI Survey Study. Am J Med Genet A. 2014 Aug;164A(8):1953-64. doi: 10.1002/ajmg.a.36584. Epub 2014 Apr 24. PMID 24764221